CLINICAL TRIAL: NCT01644032
Title: Telemedically Supported Analgesia in the Emergency Medical Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-1003-0034-3; PtJ-Az.: z0909im002b (Other Grant/Funding Number: PTJ)
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Indication for Analgesia; Emergency Medical Service; Teleconsultation
Keywords: telemedicine; teleconsultation; analgesia; emergency; prehospital
MeSH Terms: conditions — Agnosia; Emergencies | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device_ Teleconsultation (Experimental): Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. In cases of emergencies, where intravenous analgesia is necessary, if patients give informed consent the paramedics can use this system to contact a so called "tele-EMS physician" with an audio-connection to the EMS team who receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team and can delegate the application of morphine and other analgesics. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene.
  The safety, efficacy and the quality of analgesia should be compared with regular EMS.
  Interventions: Other: Teleconsultation
- Historical Control Period (No Intervention): After completion of the study arm, matched pairs from a historical phase (without the ability of teleconsultation) were searched. Local cases were always matched with comparable controls from the same location.

INTERVENTIONS:
Other: Teleconsultation — Teleconsultation between paramedics and an EMS physician
  Arms: Device_ Teleconsultation

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of telemedically supported and delegated pain therapy in the Emergency Medical Service (EMS).

DETAILED DESCRIPTION:
Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. In cases of emergencies, where intravenous analgesia is necessary, the paramedics can use this system to contact a so called "tele-EMS physician" after consent of the patient is obtained. The tele-EMS physician has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team and can delegate the application of morphine and other analgesics. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene.

All regular ambulances of the five districts are not allowed to administer analgesics without an physician on-scene. They have to call an Advanced Life Support response unit, staffed with an EMS physician, who carries out all kinds of ALS interventions.

The safety, efficacy and the quality of analgesia should be compared with regular EMS.

ELIGIBILITY:
Inclusion Criteria:

* Verbal consent obtained or patient is unable to consent due to the severity of the emergency
* Indication for analgesia

Exclusion Criteria:

* Refused consent
* No indication for analgesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Rate of complications | 2 hours
  Definition of complications: respiratory insufficiency, allergic reaction, circulatory insufficiency

SECONDARY OUTCOMES:
Pain level | average 1 hour
  Pain level measured with numerical rating scale
Incidence of nausea and vomiting | 2 hours
Time intervals | average 1 hour
  on-scene time, contact to hospital time
Medications and dosages | average 1 hour
  Evaluation and description of the used medications and dosages

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital Aachen, Germany, Department of Anesthesiology; Jörg Brokmann, Dr., Principal Investigator — University Hospital Aachen, Germany, Emergency Department
Locations (1):
- University Hospital Aachen, Aachen, Germany